CLINICAL TRIAL: NCT04412226
Title: Effect of Using Barrier Devices for Intubation in COVID-19 Patients: Randomized, Prospective, Manikin Study
Brief Title: Effect of Using Barrier Devices for Intubation in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ASIM ENES ÖZBEK, Principal Investigator, Derince Training and Research Hospital
Other Study IDs: 2020/56
Record Dates: First submitted 2020-05-31; First posted 2020-06-02 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Intubation, Intratracheal; COVID-19
Keywords: aerosol box; COVID-19; intubation; personal protective equipment; barrier device
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: aerosol box — The aerosol box is a barrier that protects the staff against the aerosols during the aerosol generating procedures like endotracheal intubation. It is a transparent cube that covers the patient's head during the endotracheal intubation. Operator can intubate the patient through the two holes for arms.
Device: transparent sheet — The transparent sheet is a barrier that protects the staff against the aerosols during the aerosol generating procedures like endotracheal intubation. It is a transparent cover that covers the patient's head and body during the endotracheal intubation. Operator can intubate the patient through the space under the cover

SUMMARY:
The aim of this study is to compare the impact of using the aerosol box and transparent sheet as an adjunct to conventional personal protective equipment on endotracheal intubation of COVID-19 patients. The effect of the head of the bed elevation will also be evaluated during the mentioned simulated scenarios.

DETAILED DESCRIPTION:
This is a randomized, prospective, manikin simulation study. Emergency medicine specialists will be participated in the study. Participants will be randomly assigned into 6 groups with a 1:1:1:1:1:1 allocation following simple randomization procedures by a program generating online random numbers. 13 participants will be recruited to the study.

Operators who will intubate the manikin will use following methods: (1) conventional personal protective equipment (PPE) with placing the manikin in the supine position. (2) aerosol box as an adjunct to PPE with placing the manikin in the supine position. (3) transparent sheet as an adjunct to PPE with placing the manikin in the supine position. (4) conventional personal protective equipment (PPE) with placing the manikin in the 30 degree the head of the bed elevated position. (5) aerosol box as an adjunct to PPE with placing the manikin in the 30 degree the head of the bed elevated position. (6) transparent sheet as an adjunct to PPE with placing the manikin in the 30 degree the head of the bed elevated position.

ELIGIBILITY:
Inclusion Criteria:

* Participants who want to participate the study

Exclusion Criteria:

* Participants who do not want to participate the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes emergency medicine specialists who wants to participate to the study.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
First pass success | 2 minutes
  Comparison of the first pass success rates for each method that were mentioned in the 'Detailed Description' of the study.

SECONDARY OUTCOMES:
Time to endotracheal intubation | 2 minutes
  The mean time to successful endotracheal intubation for each method that were mentioned in the 'Detailed Description' of the study.
Difficulty level of accessing the equipment | 2 minutes
  Grading the difficulty of accessing the equipment on a 5-point Likert scale for each method that were mentioned in the 'Detailed Description' of the study.
Difficulty level of inserting the endotracheal tube into the glottis | 2 minutes
  Grading the difficulty of inserting the endotracheal tube into the glottis on a 5-point Likert scale for each method that were mentioned in the 'Detailed Description' of the study.
Clarity of the view of the patient's face | 2 minutes
  Grading the clarity of the view of the patient's face on a 5-point Likert scale for each method that were mentioned in the 'Detailed Description' of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Derince Training and Research Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Tran K, Cimon K, Severn M, Pessoa-Silva CL, Conly J. Aerosol generating procedures and risk of transmission of acute respiratory infections to healthcare workers: a systematic review. PLoS One. 2012;7(4):e35797. doi: 10.1371/journal.pone.0035797. Epub 2012 Apr 26. PMID 22563403
- [Background] Feldman O, Meir M, Shavit D, Idelman R, Shavit I. Exposure to a Surrogate Measure of Contamination From Simulated Patients by Emergency Department Personnel Wearing Personal Protective Equipment. JAMA. 2020 May 26;323(20):2091-2093. doi: 10.1001/jama.2020.6633. PMID 32338711
- See also: Aerosol Box — http://sites.google.com/view/aerosolbox/home?authuser=0